CLINICAL TRIAL: NCT07372534
Title: Effects of Craniosacral Therapy Added to a Home Exercise Program on Pain, Heart Rate Variability, and Functional Outcomes in Patients With Gonarthrosis: A Randomized Controlled Trial
Brief Title: Efficacy of Craniosacral Therapy in Patients With Gonarthrosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Rabia Tugba Kilic, Principal Investigator, PT, PhD Candidate, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-149
Record Dates: First submitted 2025-12-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Gonarthrosis; Knee Osteoarthritis
Keywords: craniosacral therapy; knee osteoarthritis; osteoarthritis; gonarthrosis; Home Exercise Program; Randomized Controlled Trial
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups. Both groups will receive a standardized home exercise program for six weeks. In addition, the experimental group will receive craniosacral therapy once weekly for six weeks, while the control group will receive the home exercise program alone. Outcomes will be assessed at baseline and after the six-week intervention period.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Craniosacral Therapy + Home Exercise Program (Experimental): Participants in the craniosacral therapy plus home exercise (CST+HBE) group will receive one forty-minute craniosacral therapy session per week for six weeks. The standardized intervention protocol will include frontal and parietal lifting-spreading, ear pulling, temporal internal rotation, atlanto-occipital release, dural tube traction, rib lifting, and diaphragm harmonization techniques, applied according to the Frymann method. All sessions will be delivered by a physiotherapist certified in craniosacral therapy under the supervision of an osteopath (Doctor of Osteopathy, R.T.T.).
  Interventions: Other: Craniosacral Therapy; Other: Home-Based Exercise Program
- Home-Based Exercise Program (Active Comparator): All participants will follow a standardized, step-by-step home-based exercise program consisting of stretching, strengthening, and range-of-motion exercises targeting the muscles surrounding the knee joint. The program will be prescribed to be performed daily for six weeks. To enhance adherence, participants will be provided with an illustrated exercise booklet and adherence will be monitored through weekly telephone calls and exercise diaries..
  Interventions: Other: Home-Based Exercise Program

INTERVENTIONS:
Other: Craniosacral Therapy — Craniosacral therapy will be administered once weekly for six weeks by a physiotherapist certified in craniosacral therapy under the supervision of an osteopath. Each session will last forty minutes and will follow a standardized protocol including frontal and parietal lifting-spreading, ear pulling, temporal internal rotation, atlanto-occipital release, dural tube traction, rib lifting, and diaphragm harmonization techniques according to the Frymann method.
  Arms: Craniosacral Therapy + Home Exercise Program
Other: Home-Based Exercise Program — All participants will perform a standardized home-based exercise program consisting of stretching, strengthening, and range-of-motion exercises targeting the muscles surrounding the knee joint. The program will be prescribed to be performed daily for six weeks. Participants will receive an illustrated exercise booklet, and adherence will be monitored through weekly telephone calls and exercise diaries.

SUMMARY:
This randomized controlled trial was designed to investigate the effects of craniosacral therapy on pain, heart rate variability, joint stiffness, physical function, quality of life, body image, kinesiophobia, and dynamic balance in adult patients with gonarthrosis. The primary research question is whether craniosacral therapy, when added to a standard home exercise program administered by physical therapists, is more effective than a home exercise program alone.

Participants will be randomly allocated into two groups. Both groups will perform a standardized home exercise program for six weeks. In addition, the experimental group will receive craniosacral therapy once weekly for six weeks, whereas the control group will receive the home exercise program only. Outcome measures will be assessed at baseline and after the six-week intervention period to compare the effectiveness of the two treatment approaches.

DETAILED DESCRIPTION:
Gonarthrosis is a prevalent degenerative joint disease characterized by pain, joint stiffness, impaired physical function, and reduced quality of life. In addition to biomechanical impairments, individuals with gonarthrosis often experience alterations in autonomic nervous system activity, psychosocial factors such as kinesiophobia and body image disturbances, and limitations in functional mobility. While therapeutic exercise is considered a cornerstone of conservative management, complementary manual therapy approaches may provide additional benefits by targeting pain modulation and neurophysiological regulation.

Craniosacral therapy is a gentle manual therapy approach that aims to influence the craniosacral system and may contribute to pain reduction and autonomic regulation. However, evidence regarding its effectiveness as an adjunct to exercise-based rehabilitation in patients with gonarthrosis remains limited.

This randomized controlled trial was designed to investigate the effects of craniosacral therapy added to a standard home exercise program on pain, heart rate variability, joint stiffness, physical function, quality of life, body image, kinesiophobia, and dynamic balance in adult patients diagnosed with gonarthrosis. The primary objective is to determine whether the addition of craniosacral therapy to a home exercise program administered by physical therapists results in superior clinical outcomes compared with a home exercise program alone.

Eligible participants will be randomly allocated into two parallel groups. Both groups will perform a standardized home exercise program for a duration of six weeks. Participants in the experimental group will additionally receive craniosacral therapy once weekly for six weeks, whereas participants in the control group will receive the home exercise program only. All outcome assessments will be conducted at baseline and after the six-week intervention period by a physiotherapist blinded to group allocation.

The home exercise program will be prescribed and monitored by physiotherapists and will include exercises targeting knee joint mobility, muscle strength, flexibility, and functional performance. Craniosacral therapy sessions will be delivered by a trained physiotherapist following standardized clinical principles. Adherence to the exercise program will be monitored throughout the intervention period.

Outcome measures will include pain intensity, heart rate variability parameters, joint stiffness, physical function, quality of life, self-efficacy, kinesiophobia, body image perception, and functional mobility. The findings of this study are expected to contribute to the understanding of the potential role of craniosacral therapy as an adjunct to exercise-based rehabilitation in the management of gonarthrosis.

ELIGIBILITY:
Inclusion Criteria:

* Age between forty and eighty-five years
* Diagnosis of knee osteoarthritis
* Ability to understand the study procedures and provision of written informed consent

Exclusion Criteria:

* Consumption of caffeine within the last four hours or use of tobacco within the last forty-eight hours prior to assessment
* Use of alcohol or recreational drugs within the last week
* Eating within two hours before the assessment
* History of neuropathic disorders
* History of unexplained syncope episodes
* Inability to move independently
* Presence of uncontrolled medical conditions, such as cardiac (e.g., angina) or respiratory (e.g., asthma) diseases
* Presence of neurological disorders, including Parkinson's disease or multiple sclerosis
* History of vascular surgery or open knee surgery, or receipt of a knee injection within the last one month
* Presence of somatic dysfunction symptoms or musculoskeletal injuries that may interfere with assessments
* Diagnosis of pregnancy, sarcopenia, cognitive impairment, or osteoporosis
* Any medical condition affecting the autonomic nervous system or immune system, including autonomic neuropathy, pure autonomic failure, autoimmune diseases, or acquired immunodeficiency syndrome

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity Measured by Visual Analog Scale (VAS) | Time Frame: Baseline and six weeks
  Pain intensity will be measured using a ten-centimeter Visual Analog Scale (VAS), where zero indicates "no pain" and ten indicates "worst imaginable pain."
Change in Low-Frequency (LF) Power | Baseline and six weeks
  Low-Frequency (LF) Power will be assessed using the Polar H10 heart rate monitor (Polar Electro, Finland). Following a fifteen-minute seated rest period, an eight-minute supine recording will be obtained. Low-frequency (LF) power will be analyzed using the Elite HRV© application.
Change in High-Frequency (HF) Power | Baseline and six weeks
  High-Frequency (HF) Power will be assessed using the Polar H10 heart rate monitor (Polar Electro, Finland). Following a fifteen-minute seated rest period, an eight-minute supine recording will be obtained. High-frequency (HF) power will be analyzed using the Elite HRV© application.
Change in LF/HF Ratio | Baseline and six weeks
  LF/HF Ratio will be assessed using the Polar H10 heart rate monitor (Polar Electro, Finland). Following a fifteen-minute seated rest period, an eight-minute supine recording will be obtained. The LF/HF ratio will be calculated using the Elite HRV© application.
Change in SDNN | Baseline and six weeks
  Standard deviation of all normal-to-normal intervals (SDNN) will be assessed using the Polar H10 heart rate monitor (Polar Electro, Finland). Following a fifteen-minute seated rest period, an eight-minute supine recording will be obtained. The standard deviation of all normal-to-normal intervals (SDNN) will be calculated using the Elite HRV© application.
Change in RMSSD | Baseline and six weeks
  Root mean square of successive differences between normal-to-normal intervals (RMSSD) will be assessed using the Polar H10 heart rate monitor (Polar Electro, Finland). Following a fifteen-minute seated rest period, an eight-minute supine recording will be obtained. The root mean square of successive differences between normal-to-normal intervals (RMSSD) will be calculated using the Elite HRV© application.

SECONDARY OUTCOMES:
Change in Pain, Joint Stiffness, and Physical Function Assessed by WOMAC | Baseline and six weeks
  Pain, stiffness, and physical function will be evaluated using the twenty-four-item Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). Items are scored on a five-point Likert scale (0-4), with higher scores indicating worse symptoms.
Change in Health-Related Quality of Life Measured by SF-36 | Baseline and six weeks
  Quality of life will be assessed using the thirty-six-item Short Form Health Survey (SF-36), with scores ranging from zero to one hundred, where higher scores indicate better perceived health status.
Change in Self-Efficacy Measured by the Arthritis Self-Efficacy Scale | Baseline and six weeks
  Self-efficacy will be evaluated using the Arthritis Self-Efficacy Scale (ASES), which includes pain, hand/arm function, and leg/foot function subdomains.
Change in Kinesiophobia Measured by the Tampa Scale for Kinesiophobia | Baseline and six weeks
  Kinesiophobia will be measured using the Tampa Scale for Kinesiophobia (TSK), with total scores ranging from seventeen to sixty-eight. Higher scores indicate greater fear of movement.
Change in Body Image Perception Measured by the Body Image Scale | Baseline and six weeks
  Body image perception will be assessed using the Body Image Scale, a forty-item self-report questionnaire. Total scores range from 40 to 200, with higher scores indicating a more positive body image perception, which reflects better outcomes.
Change in Functional Mobility Measured by the Timed Up and Go Test | Baseline and six weeks
  Functional mobility will be evaluated using the Timed Up and Go (TUG) test. Shorter completion times indicate better functional mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27347698/